CLINICAL TRIAL: NCT05798364
Title: Household Transmission Dynamics of Multidrug Resistant Enterobacterales
Acronym: HOME
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220479
Record Dates: First submitted 2023-01-06; First posted 2023-04-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Adults Patients, With Fecal Carriage of Multi-Drug Resistant Enterobacterales (MDR-E)
Keywords: Multi-Drug Resistant Enterobacterales ; ; ; ;; Extended-Spectrum Beta-Lactamase producing Enterobacterales; Carbapenemase-Producing Enterobacterales; Transmission; Community; households; Mathematical modelling; microbiota; Whole genome sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stools samples, isolated MDR E strains
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Index patients: Adults MDR-E carriers.
- Household members: Adults or children living in the same household as the index case (i.e. sharing the same kitchen and/or bathroom and/or toilets) during the 3 months following inclusion

SUMMARY:
The HOME study will prospectively follow a cohort of Multi-Drug Resistant Enterobacterales (MDR-E) carriers after hospital discharge, and their related household members over a 3-month period. The main objective is to estimate the rate of confirmed transmissions of MDR-E from the index cases to related household members, and identify predictors associated with transmission. Transmission will be confirmed by comparing genomic analysis of the MDR-E strains isolated both in the index patient and his/her household members, based on the number of Single nucleotide polymorphisms (SNPs) differences between nearby genomes by Variant Calling. Multifactorial processes involved in MDR-E transmission in households will be explored with stochastic individual-based modelling. The parameterized model will be used to simulate and assess different strategies of control of MDR-E emergence and transmission to households. The impact of modifying patterns of human-contacts, promote hygiene and control barriers (decontamination of objects or surfaces, variations in antibiotic use, reinforcement of hand hygiene) will be assessed.

DETAILED DESCRIPTION:
Multi-Drug Resistant Enterobacterales (MDR-E), i.e. Extended-Spectrum Beta-Lactamase producing Enterobacterales (ESBL-E) and Carbapenemase-Producing Enterobacterales (CPE) are spreading worldwide. Although initially considered a healthcare-associated problem, reports of ESBL-E carriage and infections in individuals without any previous exposure to health care raise concerns on their alarming dissemination in the community. Very few reports investigated the dynamics of transmission of MDR-E from carriers to household members. Risk factors of acquisition (related to the strain, household habits, travel, occupational activities…) were poorly assessed.

Quantifying and understanding the mechanisms of household transmission is of major importance to elaborate control strategies specifically designed to the community.

The main objective is to estimate the rate of confirmed transmissions of MDR-E from an index case to related household members.

The primary endpoint is defined by the secondary attack rate (SAR) for confirmed transmissions, i.e. the proportion of confirmed (based on genetic analysis of strains) acquisitions of MDR-E in all household members over the study period (three months).

Screening of eligible patients will rely on an automated daily request of all MDR-E positive samples that is already implemented in the participating centers.

Information on the study will be given to eligible patients, those who meet eligibility criteria and willing to participate will be asked to ive non-opposition.

Seven days before hospital discharge, index patients who consent to participate will provide a fecal sample to be screened for MDR-E carriage. If the patient is still positive at discharge for MDR-E fecal carriage, he/she will be included in the cohort (=index case). His/her household members (=HH members) will then be invited to participate and included after agreement.

After inclusion, index cases and household members will be prospectively followed-up for 3 months (+/-7 days), and asked to provide self-collected stool samples and questionnaires on day7, day15, day21, day30, month2 and month3.

Self-collected stool samples will be mailed to the reference microbiology laboratory (Bichat) with self-filled questionnaires.

In addition, in the context of the ancillary study:

To obtain accurate data on interactions between household members, Ultra Wide Band (UWB) systems will be used. During 4 days, index cases and household members will wear a small wireless sensor that records continuously the identity of other sensors that are in close proximity. For each household, recording will be performed on 2 week days and 2 week-end days (Saturday and Sunday).

Proportion of transmissions in all household members over the study period (SAR) and 95% confidence intervals will be calculated at the end of follow-up for both probable and confirmed transmissions and described according to household size and index-case population type. Kaplan Meier survival analysis will be used to estimate the median time to (first) acquisition among household members and a Cox shared frailty-model to study variables associated with acquisition index-case and household members' potential exposures, household's characteristics, MDR-E abundance in index case-patients, intestinal microbiota diversity and composition). Additionally, a stochastic individual based model to capture the multifactorial processes involved in MDR-E transmission will developed. Several models of increasing complexity will be built in order to compare their likelihood given the acquisitions observed over time in the different households. The model will be integrated in an inference framework to analyse the data and estimate model parameters (eg transmission rates for the different routes). The inference techniques will involve bayesian statistics, probably Markov Chain Monte Carlo with data augmentation. The different models will be compared based on specific criterion, such as the Deviance Information Criterion (DIC). The parameterized model selected in the preceding step will be used to simulate and assess different strategies of control of MDR-E emergence and transmission to households.

ELIGIBILITY:
Inclusion criteria :

Index patients

* adults (≥ 18 years)
* hospitalized in participating hospitals
* positive for MDR-E fecal carriage on routine screening during hospital stay
* with no documented MDR-E fecal carriage in the 12 months preceding current hospitalization
* regularly living with at least two additional household members who expressed their non-opposition to participate.
* planning to live in Ile de France for the next three months Household members
* adults or children living in the same household as the index case (i.e. sharing the same kitchen and/or bathroom and/or toilets) during the 3 months following inclusion, and who expressed their non-opposition to participate.
* planning to live in Ile de France for the next three months

Exclusion criteria :

Lack of non-opposition to participate and to use clinical data

* Subject under legal protection (guardianship)
* Subject deprived of liberty under judicial constraint
* Subject undergoing psychiatric care
* Lack of affiliation to a social security scheme Secondary exclusion criteria
* Index member negative for MDR-E fecal carriage either before discharge (D-7 to D-2) or on day of discharge (D0)."

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults MDR-E carriers (index patients) and their related household members (children, pregnant and breastfeeding women included)
Sampling Method: Non-Probability Sample
Enrollment: 507 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Secondary attack rate (SAR) for confirmed transmissions, i.e. the proportion of confirmed acquisitions of MDR-E (based on genetic analysis of strains) in all household members over the study period | 3 months

SECONDARY OUTCOMES:
SAR for possible transmissions, i.e. the proportion of possible (based on phenotypic analysis of strains) acquisitions of MDR-E in all household members over the study period | 3 months
Hazard ratios of epidemiological and microbiological factors associated with confirmed transmission | 3 months
Median time to decolonization in MDR-E carriers (index or household members) | 3 months
Hazard ratios of epidemiological and microbiological factors associated with decolonization | 3 months
Diversity indices of the microbiota (Shannon diversity index) in pairs index/household member with or without confirmed transmission | 3 months
Number of interactions between index patients and household participants | 4 days
Duration of interactions between index and household participants | 4 days
Number of observed Operational Taxonomic Units in pairs index/household member with or without confirmed transmission | 3 months
Bray-Curtis unweighted UniFrac distance in pairs index/household member with or without confirmed transmission | 3 months
Bray-Curtis dissimilarity in pairs index/household member with or without confirmed transmission | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kernéis Solen, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat Hospital, Paris, Île-de-France Region, France